CLINICAL TRIAL: NCT04803305
Title: A 6-WEEK, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN STUDY TO ASSESS THE EFFECT OF REPEATED SUBCUTANEOUS ADMINISTRATION OF PF-06946860 ON APPETITE IN PARTICIPANTS WITH ADVANCED CANCER AND ANOREXIA, FOLLOWED BY AN 18-WEEK OPEN-LABEL TREATMENT PERIOD
Brief Title: Study to Compare the Effects of Repeated Doses of an Investigational New Drug and a Placebo on Appetite in Advanced Cancer and Anorexia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C3651010
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer; Prostate Cancer; Breast Cancer; Ovarian Cancer; Loss of Appetite; Fatigue; Cachexia; Anorexia
Keywords: cancer, anorexia, cachexia, weight loss, loss of appetite, fatigue
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Anorexia; Fatigue; Cachexia; Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, sponsor open for 6-week double-blind treatment period followed by an optional 18-week open-label treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-Blind PF-06946860 Treatment followed by Open Label PF-06946860 Treatment (Experimental): subcutaneous injection
  Interventions: Drug: PF-06946860
- Double-Blind Placebo Treatment followed by Open-Label PF-06946860 Treatment (Placebo Comparator): subcutaneous injection
  Interventions: Drug: PF-06946860; Drug: Placebo for PF-06946860

INTERVENTIONS:
Drug: PF-06946860 — subcutaneous injection
Drug: Placebo for PF-06946860 — subcutaneous injection
  Arms: Double-Blind Placebo Treatment followed by Open-Label PF-06946860 Treatment

SUMMARY:
Study to compare the effects of the investigational new drug (PF-06946860) and a placebo on appetite and to find out how participants with advanced cancer and anorexia feel after receiving repeated subcutaneous (SC-injected under the skin) doses.

DETAILED DESCRIPTION:
A 6 week double blind study to compare the effects of the investigational new drug (PF-06946860) and a placebo on appetite and to find out how participants with advanced cancer and anorexia feel after receiving repeated doses injected under the skin (subcutaneously).

During the initial 6-week treatment period (Part A), a total of 2 doses of study drug or placebo will be administered 3 weeks apart. Each dose contains two injections. Part B is an optional 18-week open-label treatment period where up to 7 doses of study drug may be administered. Part B does not include placebo.

Assessments include:

* Measure the impact of the study drug on appetite, fatigue, and pain questionnaires
* Body weight measurements
* Blood samples to evaluate safety and additional endpoints including the amount of the study drug in the blood and the effects of the study drug on levels of a specific cytokine.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of non-small cell lung, pancreatic, colorectal, prostate, breast or ovarian cancer which, in the treating oncologist's assessment, is considered advanced.
* Anorexia as defined by a score of ≤5 in the Cancer-Related Cachexia Symptom Assessment Appetite 7-day recall scale
* Meets any of the following criteria at Randomization:

  * Not currently receiving antineoplastic therapy
  * On standard of care systemic antineoplastic therapy or treatment without curative intent
* Signed informed consent.

Key Exclusion Criteria:

* Receiving tube feedings or parenteral nutrition at the time of Screening or Randomization.
* Current active reversible causes of decreased food intake.
* Current, severe gastrointestinal disease
* Participants with known symptomatic brain metastases requiring steroids.
* Active uncontrolled bacterial, fungal, or viral infection, including HBV, HCV, HIV or participants with known AIDS-related illness
* inadequate renal or liver function.
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (32):
  - CARTI Cancer Center, Little Rock, Arkansas
  - Tower Hematology Oncology Medical Group (THO), Beverly Hills, California
  - Ventura County Hematology- Oncology Specialists, Camarillo, California
  - Cedars- Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Providence Medical Foundation, Santa Rosa, California
  - Ventura County Hematology-Oncology Specialists, Ventura, California
  - Lutheran Medical Center, Wheat Ridge, Colorado
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Bozeman Health Cancer Center, Bozeman, Montana
  - Bozeman Health Deaconess Hospital d/b/a Bozeman Health Clinical Research, Bozeman, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology-Paris, Paris, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Cancer Center IDS Pharmacy, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - UVA Health System; Attention: GI Team, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - MultiCare Regional Cancer Center - Gig Harbor Medical Park, Gig Harbor, Washington
  - Moses Lake Clinic, Moses Lake, Washington
  - MultiCare Regional Cancer Center - Puyallup, Puyallup, Washington
  - Medical Oncology Associates, PS (dba Summit Cancer Centers), Spokane Valley, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington
  - Wenatchee Valley Hospital, Wenatchee, Washington
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were enrolled into the study and treated.
Groups:
- Placebo -> OL PF-06946860 200mg Q3W: Participants received placebo during the 6-week double-blind phase (Part A) 3 weeks apart (Q3W) subcutaneously (SC). Starting at the Week 6 visit, participants who continued to the optional open-label treatment (OLT) period of up to 18 weeks (Part B) had an opportunity to receive up to 7 additional doses of PF-06946860 200 mg Q3W. Each dose was comprised of two 1 mL SC injections which were administered consecutively.
- PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W: Participants received PF-06946860 200 mg during the 6-week double-blind phase (Part A) Q3W SC. Starting at the Week 6 visit, participants who continued to the optional OLT period of up to 18 weeks (Part B) had an opportunity to receive up to 7 additional doses of PF-06946860 200 mg Q3W. Each dose was comprised of two 1 mL SC injections which were administered consecutively.
Period: Part A: 6-week Double-blind Treatment
Arm/Group | Placebo -> OL PF-06946860 200mg Q3W | PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W
Started | 6 | 12
Completed | 5 | 9
Not Completed | 1 | 3
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0
Period: Part B: OLT Period up to 18 Weeks
Arm/Group | Placebo -> OL PF-06946860 200mg Q3W | PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W
Started | 5 | 9
Completed | 2 | 5
Not Completed | 3 | 4
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Death | 1 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Placebo -> OL PF-06946860 200mg Q3W: Participants received placebo during the 6-week double-blind phase (Part A) Q3W SC. Starting at the Week 6 visit, participants who continued to the optional OLT period of up to 18 weeks (Part B) had an opportunity to receive up to 7 additional doses of PF-06946860 200 mg Q3W. Each dose was comprised of two 1 mL SC injections which were administered consecutively.
- Total: Total of all reporting groups
Arm/Group | Placebo -> OL PF-06946860 200mg Q3W | PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.95) | 74.0 (9.12) | 72.0 (8.99)
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0
  18-44 | 0 | 0 | 0
  45-64 | 2 | 2 | 4
  >=65 | 4 | 10 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 11 | 16
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 11 | 14
  Black or African American | 3 | 0 | 3
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cancer-Related Cachexia Symptom Assessment in Appetite Score at Week 4 in Part A
Description: The Cancer-Related Cachexia Symptom Assessment-Appetite was a self-reported questionnaire that measured the severity of anorexia. The measure consisted of 1 question that asked study participants to rate their appetite over the past 7 days from 0-"no appetite" to 10-"very good appetite", where higher score indicated better appetite.
  In this Outcome Measure (OM), changes from baseline in the Cancer-Related Cachexia Symptom Assessment-Appetite score at Week 4 were summarized descriptively by treatment group.
Time Frame: Baseline, Week 4
Population: The analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. The number analyzed in each group was the number of participants with non-missing data in the analysis set at a given visit. Number of participants analyzed/number analyzed = number of participants evaluable for this OM in each treatment group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a Scale
Groups:
- Placebo: Participants received placebo during the 6-week double-blind phase (Part A) Q3W SC.
- PF-06946860 200mg Q3W: Participants received PF-06946860 200 mg during the 6-week double-blind phase (Part A) Q3W SC.
Arm/Group | Placebo | PF-06946860 200mg Q3W
Number analyzed (Participants) | 5 | 9
Units on a Scale | 2.45 [1.01 to 3.88] | 1.84 [0.79 to 2.90]
Statistical Analysis 1: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = -0.60, 90% CI 2-sided [-2.38 to 1.18], Standard Error of Mean 1.01 — Week 4

2. Secondary Outcome: Change From Baseline in Cancer-Related Cachexia Symptom Assessment in Appetite Score at Weeks 1, 2, 3, 5 and 6 in Part A
Description: The Cancer-Related Cachexia Symptom Assessment-Appetite was a self-reported questionnaire that measured the severity of anorexia. The measure consisted of 1 question that asked study participants to rate their appetite over the past 7 days from 0-"no appetite" to 10-"very good appetite", where higher score indicated better appetite.
  In this OM, changes from baseline in the Cancer-Related Cachexia Symptom Assessment-Appetite score were summarized descriptively by treatment group and timepoint.
Time Frame: Baseline, Weeks 1, 2, 3, 5 and 6
Population: The analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. The number analyzed at each timepoint in each group was the number of participants with non-missing data in the analysis set at a given visit. Number of participants analyzed = number of participants evaluable for this OM, number analyzed = number of participants evaluable at each timepoint for each treatment group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | PF-06946860 200mg Q3W
Number analyzed (Participants) | 6 | 12
Units on a Scale
  Week 1: number analyzed (Participants) | 3 | 8
  Week 1 | 0.99 [-0.66 to 2.64] | 2.19 [1.17 to 3.20]
  Week 2: number analyzed (Participants) | 4 | 9
  Week 2 | 1.11 [-0.03 to 2.25] | 2.21 [1.45 to 2.98]
  Week 3: number analyzed (Participants) | 5 | 11
  Week 3 | 1.27 [-0.35 to 2.89] | 2.30 [1.20 to 3.41]
  Week 5: number analyzed (Participants) | 4 | 9
  Week 5 | 1.95 [0.27 to 3.63] | 1.95 [0.82 to 3.08]
  Week 6: number analyzed (Participants) | 4 | 9
  Week 6 | 2.41 [0.49 to 4.33] | 1.61 [0.32 to 2.90]
Statistical Analysis 1: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 1.20, 90% CI 2-sided [-0.75 to 3.15], Standard Error of Mean 1.07 — Week 1
Statistical Analysis 2: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 1.10, 90% CI 2-sided [-0.28 to 2.49], Standard Error of Mean 0.78 — Week 2
Statistical Analysis 3: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 1.03, 90% CI 2-sided [-0.93 to 2.99], Standard Error of Mean 1.11 — Week 3
Statistical Analysis 4: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-2.02 to 2.02], Standard Error of Mean 1.14 — Week 5
Statistical Analysis 5: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = -0.80, 90% CI 2-sided [-3.11 to 1.51], Standard Error of Mean 1.29 — Week 6

3. Secondary Outcome: Change From Baseline in Cancer-Related Cachexia Symptom Assessment in Fatigue Score at Weeks 1, 2, 3, 4, 5 and 6 in Part A
Description: The Cancer-Related Cachexia Symptom Assessment-Fatigue was a self-reported questionnaire that measured the severity of fatigue. The measure consisted of 1 question that asked study participants to rate their fatigue over the past 7 days from 0-"no fatigue" to 10-"worst possible fatigue", where higher score indicated worse fatigue.
  In this OM, changes from baseline in the Cancer-Related Cachexia Symptom Assessment-Fatigue score were summarized descriptively by treatment group and timepoint.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | PF-06946860 200mg Q3W
Number analyzed (Participants) | 6 | 12
Units on a Scale
  Week 1: number analyzed (Participants) | 3 | 8
  Week 1 | 1.84 [-1.47 to 5.16] | 1.52 [-0.57 to 3.60]
  Week 2: number analyzed (Participants) | 4 | 9
  Week 2 | 0.04 [-2.71 to 2.80] | -2.12 [-3.91 to -0.34]
  Week 3: number analyzed (Participants) | 5 | 11
  Week 3 | -1.21 [-2.33 to -0.09] | -0.49 [-1.23 to 0.25]
  Week 4: number analyzed (Participants) | 5 | 9
  Week 4 | -1.00 [-2.40 to 0.40] | -0.55 [-1.57 to 0.48]
  Week 5: number analyzed (Participants) | 4 | 9
  Week 5 | -0.92 [-2.47 to 0.63] | -0.24 [-1.31 to 0.82]
  Week 6: number analyzed (Participants) | 4 | 9
  Week 6 | -1.13 [-2.40 to 0.15] | 0.74 [-0.09 to 1.57]
Statistical Analysis 1: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = -0.32, 90% CI 2-sided [-4.18 to 3.53], Standard Error of Mean 1.98 — Week 1
Statistical Analysis 2: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = -2.16, 90% CI 2-sided [-5.49 to 1.16], Standard Error of Mean 1.58 — Week 2
Statistical Analysis 3: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 0.72, 90% CI 2-sided [-0.62 to 2.06], Standard Error of Mean 0.76 — Week 3
Statistical Analysis 4: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 0.45, 90% CI 2-sided [-1.29 to 2.20], Standard Error of Mean 0.97 — Week 4
Statistical Analysis 5: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 0.68, 90% CI 2-sided [-1.21 to 2.57], Standard Error of Mean 1.04 — Week 5
Statistical Analysis 6: Comparison: Placebo vs PF-06946860 200mg Q3W; Test type: Superiority; Mean Difference (Final Values) = 1.86, 90% CI 2-sided [0.34 to 3.39], Standard Error of Mean 0.84 — Week 6

4. Secondary Outcome: Number of Participants With All-Causality Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in Part A
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs are events between first dose of study drug and up to discharge from study that are absent before treatment or that worsen relative to pretreatment state. An SAE is any untoward medical occurrence at any dose that: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect.
Time Frame: Day 1 through Week 6 (for a period of 6 weeks)
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06946860 200mg Q3W
Number analyzed (Participants) | 6 | 12
Participants
  Participants With All-Causality TEAEs | 4 | 7
  Participants With All-Causality SAEs | 1 | 3

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities in Part A
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, erythrocytes, erythrocytes mean corpuscular volume, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular hemoglobin concentration, platelets, leukocytes, lymphocytes, basophils, eosinophils and monocytes), chemistry (bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, blood urea nitrogen, creatinine, urate, sodium, potassium, chloride, calcium, bicarbonate and glucose) and urine (pH, urine glucose, ketones, urine protein, urine hemoglobin, urobilinogen, urine bilirubin, nitrite, leukocyte esterase, urine erythrocytes [/high power field (HPF)], urine leukocytes [/HPF] and hyaline casts [/low power field (LPF)]).
Time Frame: Days 1, 22 and 43
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention, with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Groups:
- PF- 06946860 200mg Q3W: Participants received PF-06946860 200 mg during the 6-week double-blind phase (Part A) Q3W SC.
Arm/Group | Placebo | PF- 06946860 200mg Q3W
Number analyzed (Participants) | 5 | 11
Participants
  Hemoglobin <0.8 x lower limit of normal (LLN) | 2 | 4
  Hematocrit <0.8 x LLN | 2 | 3
  Erythrocytes <0.8 x LLN | 1 | 4
  Erythrocytes Mean Corpuscular Volume <0.9 x LLN | 0 | 0
  Erythrocytes Mean Corpuscular Volume >1.1 x upper limit of normal (ULN) | 0 | 1
  Erythrocytes Mean Corpuscular Hemoglobin <0.9 x LLN | 0 | 1
  Erythrocytes Mean Corpuscular Hemoglobin >1.1 x ULN | 0 | 0
  Erythrocytes Mean Corpuscular Hemoglobin Concentration <0.9 x LLN | 0 | 0
  Erythrocytes Mean Corpuscular Hemoglobin Concentration >1.1 x ULN | 0 | 0
  Platelets <0.5 x LLN | 0 | 0
  Platelets >1.75 x ULN | 0 | 1
  Leukocytes <0.6 x LLN | 1 | 0
  Leukocytes >1.5 x ULN | 0 | 0
  Lymphocytes <0.8 x LLN | 2 | 6
  Lymphocytes >1.2 x ULN | 0 | 0
  Basophils >1.2 x ULN | 0 | 1
  Eosinophils >1.2 x ULN | 0 | 0
  Monocytes >1.2 x ULN | 0 | 1
  Bilirubin >1.5 x ULN | 0 | 0
  Aspartate Aminotransferase >3.0 x ULN | 0 | 0
  Alanine Aminotransferase >3.0 x ULN | 0 | 0
  Alkaline Phosphatase >3.0 x ULN | 0 | 2
  Protein <0.8 x LLN | 1 | 0
  Protein >1.2 x ULN | 0 | 0
  Albumin <0.8 x LLN | 0 | 0
  Albumin >1.2 x ULN | 0 | 0
  Blood Urea Nitrogen >1.3 x ULN | 0 | 0
  Creatinine >1.3 x ULN | 0 | 1
  Urate >1.2 x ULN | 0 | 0
  Sodium <0.95 x LLN | 0 | 0
  Sodium >1.05 x ULN | 0 | 0
  Potassium <0.9 x LLN | 0 | 0
  Potassium >1.1 x ULN | 0 | 0
  Chloride <0.9 x LLN | 0 | 0
  Chloride >1.1 x ULN | 0 | 0
  Calcium <0.9 x LLN | 0 | 0
  Calcium >1.1 x ULN | 0 | 0
  Bicarbonate <0.9 x LLN | 1 | 1
  Bicarbonate >1.1 x ULN | 0 | 0
  Glucose <0.6 x LLN | 0 | 0
  Glucose >1.5 x ULN | 1 | 2
  pH <4.5 | 0 | 0
  pH >8 | 0 | 0
  Urine Glucose >=1 | 0 | 1
  Ketones >=1 | 0 | 0
  Urine Protein >=1 | 2 | 0
  Urine Hemoglobin >=1 | 0 | 2
  Urobilinogen >=1 | 0 | 0
  Urine Bilirubin >=1 | 0 | 0
  Nitrite >=1 | 0 | 1
  Leukocyte Esterase >=1 | 1 | 2
  Urine Erythrocytes (/HPF) >=20: number analyzed (Participants) | 2 | 4
  Urine Erythrocytes (/HPF) >=20 | 0 | 1
  Urine Leukocytes (/HPF) >=20: number analyzed (Participants) | 3 | 6
  Urine Leukocytes (/HPF) >=20 | 0 | 1
  Hyaline Casts (/LPF) >1: number analyzed (Participants) | 0 | 2
  Hyaline Casts (/LPF) >1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Part A: Day 1 through Week 6 Part A + Part B: up to 24 weeks
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
  AE data was planned to be collected and analyzed separately for Part A and Part A + Part B combined. No individual AE analysis was done for Part B.
Arm/Group | Placebo | PF-06946860 200mg Q3W | Placebo -> OL PF-06946860 200mg Q3W | PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W
All-Cause Mortality (participants affected / at risk) | 1/6 | 2/12 | 2/6 | 4/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/12 | 2/6 | 5/12
Other Adverse Events (participants affected / at risk) | 4/6 | 4/12 | 6/6 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | PF-06946860 200mg Q3W (N=12) | Placebo -> OL PF-06946860 200mg Q3W (N=6) | PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W (N=12)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | PF-06946860 200mg Q3W (N=12) | Placebo -> OL PF-06946860 200mg Q3W (N=6) | PF-06946860 200mg Q3W -> OL PF-06946860 200mg Q3W (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT04803305/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT04803305/SAP_001.pdf